CLINICAL TRIAL: NCT02642250
Title: Chemical, Biological and Comparative Clinical Evaluation of Entoban to Determine Safety and Efficacy for the Treatment of Chronic Diarrhea
Brief Title: Comparative Evaluation of Herbal and Allopathic Drugs for the Treatment of Chronic Diarrhea
Acronym: HA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shifa Ul Mulk Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hafiz Muhammad Asif, Sadia Shakeel, Shifa Ul Mulk Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Entb-1117
Record Dates: First submitted 2015-12-12; First posted 2015-12-30 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Diarrhea
Keywords: safety; efficacy
MeSH Terms: interventions — Metronidazole; Entoban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entoban Capsules (Experimental): Entoban is the combination of Holarrhena antidysenterica, Berberis aristata, Symplocos racemosa, Querecus infectoria and Helicteres isora.
  Interventions: Drug: Entoban
- Metronidazole DS (Experimental): Metronidazole DS(400 mg) is commonly used to treat diarrhea.It eliminates bacteria and other microorganisms that cause infections of the reproductive system, gastrointestinal tract, skin, vagina, and other areas of the body.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — The data will be recorded for physical examination including gender , age, height, weight, temperature, heart rate ,respiratory rate and blood pressure of the subject, number of stool per day, stool with or without mucus or mixed with blood along with abdominal cramps, dehydration, nausea, vomiting and related clinical information will be carefully recorded. Statistical tools and tabulated results will be used to identify the similarities and differences in safety, efficacy and tolerability of treatment.
  Arms: Metronidazole DS
Drug: Entoban — To evaluate the safety and efficacy of coded herbal formulation (Entoban) through randomized clinical study and compared with Metronidazole DS for treatment of gastrointestinal infections for improving the health of the community with due regard to the prevalence of disease and the feasibility of using alternative treatments.
  Arms: Entoban Capsules

SUMMARY:
Revival of significance and the emergent market of herbal medicinal products necessitate strong commitment by the stakeholders to safeguard the end users. The variability in the concentrations of constituents of plant material, coupled with the variety of extraction techniques and processing steps used by different manufacturers, results in distinct inconsistency in the quality of herbal products. The present study will be directed to a polyherbal formulation Entoban which integrates an outstanding blend of herbs that have been used for decades to eradicate microorganisms and worms from gastrointestinal tract. It is the combination of Holarrhena antidysenterica, Berberis aristata, Symplocos racemosa, Querecus infectoria and Helicteres isora. The current study would target the chemical assessment, pharmacological and comparative clinical evaluation of Entoban to assure its safety and efficacy.

DETAILED DESCRIPTION:
The study will be adopted to compare the efficacy, tolerability, and safety of Entoban using Metronidazole DS as a comparator. The study was carried out in XYZ hospital from Jan 2015 to Dec 2015. The participants will be selected on the basis of inclusion and exclusive criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults between the age of 18-60 years who were suffering from diarrhea of presumed infectious origin and willing to participate were eligible for inclusion in the study.

Exclusion Criteria:

* Exclusion criteria were the presence of chronic
* Iatrogenic, or bloody diarrhea, having received antibiotic treatment for other medical or surgical problems
* Having a history of renal or hepatic dysfunction
* Having a concomitant infection.
* Patients receiving treatment with an anti-diarrheal drug in the five days prior to the study were also excluded.
* Pregnant or lactating women and women planning pregnancy were also ineligible for study participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Stool D/R | 5 days
  The primary efficacy criterion will be the frequency and consistency of diarrhea in hours, from the first treatment dose to recovery. It will be evaluated through stool D/R. Stool D/R described the consistency, frequency and other important features of stool. Semisolid stool consistency with 1-2/day will be considered significant.

SECONDARY OUTCOMES:
Improvement in clinical symptoms such as abdominal pain, abdominal distension, etc will be secondary outcome measures | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Khan Usman Ghani, Ph. D, Study Director — Hamdard University Karachi
Locations (1):
- Shifa Ul MUlk Memorial Hospital, Karachi, Pakistan

REFERENCES:
- [Derived] Shakeel S, Usmanghani K, Asif HM. Efficacy and safety of Entoban for the treatment of chronic diarrhea. Pak J Pharm Sci. 2016 Nov;29(6 Suppl):2349-2353. PMID 28167477